CLINICAL TRIAL: NCT02193750
Title: Assessing the Tolerability of Oligosaccharide Supplementation in Patients With Crohn's Disease: A Randomized, Controlled Trial
Brief Title: Assessing the Tolerability of Oligosaccharide Supplementation in Patients With Crohn's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The team decided to close this study since we are not recruiting and collecting any data.
Sponsor: University of British Columbia (Other)
Collaborators: The Alfred (Other); Melbourne Health (Other)
Responsible Party: Principal Investigator, Brian Bressler, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: H14-01420
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 1 placebo muesli bars and 1 serving placebo muesli per day (0.55 g total fructans/GOS)
  Interventions: Dietary Supplement: Placebo
- Moderate Oligosaccharide Group (Experimental): 1 placebo muesli bar and 1 serving intervention muesli per day (3.25 g total fructans/GOS)
  Interventions: Dietary Supplement: Moderate Oligosaccharide Group
- High Oligosaccharide Group (Experimental): 1 intervention muesli bar and 1 serving intervention muesli per day (5.43 total fructans/GOS)
  Interventions: Dietary Supplement: High Oligosaccharide Group

INTERVENTIONS:
Dietary Supplement: Placebo — 1 placebo muesli bar and 1 serving placebo muesli per day (0.55 g total fructans/GOS)
  Arms: Placebo
Dietary Supplement: Moderate Oligosaccharide Group — 1 placebo muesli bar and 1 serving intervention muesli per day (3.25 g total fructans/GOS)
  Arms: Moderate Oligosaccharide Group
Dietary Supplement: High Oligosaccharide Group — 1 placebo muesli bar and 1 serving placebo muesli per day (5.43 g total fructans/GOS)
  Arms: High Oligosaccharide Group

SUMMARY:
The investigators hypothesize that a novel method for oligosaccharide supplementation, in the form of nutritional bars and/or muesli high in fructans and galacto-oligosaccharides (GOS), will be a safe and tolerable therapeutic intervention in patients with Crohn's disease (CD) in remission.

DETAILED DESCRIPTION:
Subjects age >/= 19 years with the diagnosis of CD for >/= 6 months, currently in remission based on the Harvey-Bradshaw Index score (</=4 points) and C-reactive protein (<5 mg/L) will be recruited from two academic hospitals and affiliated gastroenterology outpatient clinics (St. Paul's Hospital, Vancouver, British Columbia, Canada; Alfred Hospital, Melbourne, Victoria, Australia).

The study is a randomized, double-blind, placebo-controlled trial that consist of a 2-week run-in period followed by a 4-week study period. Prior to study entry, a screening visit will be required for all potential participants. If a participant meets the inclusion criteria, they will be randomized to either a placebo (0.55 g total fructans/GOS), a moderate oligosaccharide group (3.25 g total fructans/GOS) or a high oligosaccharide group (5.43 g total fructans/GOS) through a computed-generated scheme within each respective center. During the run-in period, enrolled subjects will undergo the following: 1) Laboratory analyses (CBC, routine biochemistry, CRP and fecal calprotectin); 2) Stool collection for fecal calprotectin analysis; 3) tolerability assessment including overall gastrointestinal symptoms and specific symptoms (abdominal bloating, abdominal pain, gut rumbling, flatulence) utilizing a 100mm visual analogue scale (VAS, 0 = no symptoms; 100 = worst symptoms ever experienced); 4) fatigue assessment utilizing a multi-dimensional fatigue impact scale (FIS); 5) health-related quality of life (HRQOL) assessment utilizing the Short Form 36-Item Health Survey (SF-36) and 6) Mood assessment utilizing the Spielberger State-Trait Personality Inventory (STPI). Participants will also meet with a registered dietitian to quantify baseline oligosaccharide consumption by completing a prospective 5-day diet diary alongside a validated food frequency questionnaire (FFQ), the Monash University Comprehensive Nutritional Assessment Questionnaire (CNAQ) that assesses oligosaccharide intake in addition to the usual nutrients [49]. Once the initial dietary assessment is complete, participants will begin up-titration of their oligosaccharide supplementation in a step-wise fashion until they reach their required daily amounts defined by their treatment group allocation. Once this is achieved, they will enter the 4 weeks of treatment or at time of relapse. Participants will undergo re-assessment during the study period at 2 weeks (Visit #3), and at study completion (Visit #4).

If a participant undergoes a CD flare during the run-in period, they will be withdrawn from the study. The end point of the study will be at 4 weeks of treatment or at time of relapse.

ELIGIBILITY:
Inclusion Criteria:

* age >/= 19 years
* diagnosed with CD for >/= 6 months, currently in remission based on the Harvey-Bradshaw Index score (</= 4 points) and C-reactive protein (<5mg/L)

Exclusion Criteria:

* unable to provide informed consent;
* have significant hepatic, renal, endocrine, respiratory, neurological, or cardiovascular disease;
* confirmed diagnosis of celiac disease, or have suspected celiac disease and are following a gluten-free diet to manage symptoms with an elevated screening anti-tissue transglutaminase antibody test;
* significant complications of CD which includes a history of extensive colonic resection, including subtotal or total colectomy, history of >/= 3 small bowel resections or received a diagnosis of short bowel syndrome, current ileostomy, colostomy or ileal-anal pouch, or a fixed symptomatic intestinal stenosis;
* antibiotic use in the 4 weeks prior to study start;
* use of any rectal preparations in the 2 weeks prior to study start;
* use of any non-steroidal anti-inflammatory drugs in the 2 weeks prior to study start;
* use of commercial probiotic supplements in the 4 weeks prior to study start
* change in CD therapy in the 4 weeks prior to study start (excluding steroid taper, however steroid dosing must be stable for 2 weeks prior to study start);
* recently been adhering to a novel dietary intervention for alternative health issues within the last 4 weeks prior to study start.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Difference in overall GI symptoms | 5 days
  The primary outcome will be the difference in overall gastrointestinal symptoms quantified by the VAS, at study completion compared to baseline, averaged over the 5-days in which the diet diaries are being completed among the 3 study groups.

SECONDARY OUTCOMES:
Tolerability assessment including overall gastrointestinal symptoms and specific symptoms | 4 weeks
  Secondary outcomes concerning tolerability will include differences in the individual gastrointestinal symptoms (abdominal bloating, abdominal pain, gut rumbling, flatulence) quantified by the VAS at study completion compared to baseline, averaged over the 5-days in which the diet diaries are being completed among the 3 study groups.
Fatigue assessment | 4 weeks
  Secondary endpoints concerning differences in the scores of the overall FIS (fatigue impact scale) and sub-categories (physical, cognitive, psychosocial) at study completion compared to baseline in all 3 study groups
Quality of Life Assessment | 4 weeks
  Secondary endpoints concerning differences in physical components summary (PCS) and the mental component summary (MSC) scores at study completion compared to baseline in all 3 study groups respectively
Mood Assessment | 4 weeks
  Secondary endpoints concerning mood that will include differences in state anxiety, state curiosity, state anger, and state depression scores of the STPI at study completion compared to baseline in all 3 study groups respectively
Disease Activity Asessment | 4 weeks
  The proportion of participants who relapse, as well as the time to relapse at study completion between groups.
Adherence Assessment | 4 weeks
  Adherence will be estimated and compared between groups at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bressler, MD, Principal Investigator — Division of Gastroenterology, Department of Medicine St. Paul's Hospital, Vancouver, BC Cananda; Peter Gibson, MD, Principal Investigator — Department of Gastroenterology Alfred Hospital, Melbourne, Australia
Locations (2):
- Department of Gastroenterology Alfred Hospital, Melbourne, Australia
- GI Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Talley NJ, Abreu MT, Achkar JP, Bernstein CN, Dubinsky MC, Hanauer SB, Kane SV, Sandborn WJ, Ullman TA, Moayyedi P; American College of Gastroenterology IBD Task Force. An evidence-based systematic review on medical therapies for inflammatory bowel disease. Am J Gastroenterol. 2011 Apr;106 Suppl 1:S2-25; quiz S26. doi: 10.1038/ajg.2011.58. No abstract available. PMID 21472012
- [Result] Kappelman MD, Rifas-Shiman SL, Kleinman K, Ollendorf D, Bousvaros A, Grand RJ, Finkelstein JA. The prevalence and geographic distribution of Crohn's disease and ulcerative colitis in the United States. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1424-9. doi: 10.1016/j.cgh.2007.07.012. Epub 2007 Sep 29. PMID 17904915
- [Result] Herrinton LJ, Liu L, Lewis JD, Griffin PM, Allison J. Incidence and prevalence of inflammatory bowel disease in a Northern California managed care organization, 1996-2002. Am J Gastroenterol. 2008 Aug;103(8):1998-2006. doi: 10.1111/j.1572-0241.2008.01960.x. PMID 18796097
- [Result] Lichtenstein GR, Hanauer SB, Sandborn WJ; Practice Parameters Committee of American College of Gastroenterology. Management of Crohn's disease in adults. Am J Gastroenterol. 2009 Feb;104(2):465-83; quiz 464, 484. doi: 10.1038/ajg.2008.168. Epub 2009 Jan 6. PMID 19174807
- [Result] Pai CG, Khandige GK. Is Crohn's disease rare in India? Indian J Gastroenterol. 2000 Jan-Mar;19(1):17-20. PMID 10659482
- [Result] El Mouzan MI, Abdullah AM, Al Habbal MT. Epidemiology of juvenile-onset inflammatory bowel disease in central Saudi Arabia. J Trop Pediatr. 2006 Feb;52(1):69-71. doi: 10.1093/tropej/fmi039. Epub 2005 Jun 9. PMID 15947013
- [Result] Ouyang Q, Tandon R, Goh KL, Ooi CJ, Ogata H, Fiocchi C. The emergence of inflammatory bowel disease in the Asian Pacific region. Curr Opin Gastroenterol. 2005 Jul;21(4):408-13. PMID 15930979
- [Result] Aghazadeh R, Zali MR, Bahari A, Amin K, Ghahghaie F, Firouzi F. Inflammatory bowel disease in Iran: a review of 457 cases. J Gastroenterol Hepatol. 2005 Nov;20(11):1691-5. doi: 10.1111/j.1440-1746.2005.03905.x. PMID 16246187
- [Result] Wright JP, Froggatt J, O'Keefe EA, Ackerman S, Watermeyer S, Louw J, Adams G, Girdwood AH, Burns DG, Marks IN. The epidemiology of inflammatory bowel disease in Cape Town 1980-1984. S Afr Med J. 1986 Jul 5;70(1):10-5. PMID 3726680